CLINICAL TRIAL: NCT07158255
Title: Effect of Exercise Training on Pain, Range of Motion, Functionality and Shoulder Architecture in Patients With Adhesive Capsulitis
Brief Title: Effects of Exercise on Adhesive Capsulitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuğba GÖNEN, Assist. Prof. Dr., Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/097
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Adhesive Capsulitis; Exercise; Ultrasonography
Keywords: adhezsiv capsulitis; pain; range of motion; functionality; shoulder architecture; exercise
MeSH Terms: conditions — Bursitis; Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants were divided into two groups. Two different interventions were administered to each group. One group will receive electrotherapy and exercise therapy. The other group will receive electrotherapy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training group (Experimental): Patients in the study group will receive 15 sessions of exercise training (daily for 3 weeks). Exercise training includes programs to increase joint range of motion and mobility at the pain threshold and to restore functionality.
  Interventions: Other: Exercise training
- Control group (Active Comparator): Patients in the control group will receive 15 sessions of electrotherapy treatment (TENS, US, Hotpack)
  Interventions: Other: electrotherapy treatment

INTERVENTIONS:
Other: electrotherapy treatment — Patients in the electrotherapy group will receive 15 sessions of TENS, hotpack, and ultrasound, 45 minutes each, 5 days a week, for 3 weeks. The treatment program is planned for 20 minutes of TENS, 15 minutes of hotpack, and 10 minutes of ultrasound.
  Arms: Control group
Other: Exercise training — In addition to electrotherapy, the patients in the study group will receive 15 sessions (45 minutes, 5 days a week, for 3 weeks) of exercise training consistent with the literature. Exercise training includes programs to increase joint range of motion and mobility at the pain threshold and to restore functionality. Following electrotherapy, upper extremity normal range of motion exercises, anterior and posterior capsule stretching exercises, pendulum exercises, wand exercises, isometric training in 3 planes, and isotonic strengthening exercises will be applied. Five exercises will be selected each day, performed under the supervision of a physiotherapist. A 2-minute rest period will be provided after each exercise, followed by a transition to the next exercise. Care will be taken to perform the exercises within the pain threshold and to ensure that the pain does not exceed a VAS score of 2.
  Arms: Exercise training group

SUMMARY:
Our study aims to investigate the effects of exercise training on pain, range of motion, functionality and shoulder architecture in patients with adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive capsulitis (AC) is a common shoulder condition characterized by a gradual increase in spontaneous pain and a limitation in glenohumeral joint range of motion. Its pathophysiology, a pathological process of capsular fibrosis following synovial inflammation, is relatively well understood, but its cause remains unknown. The literature on the treatment of frozen shoulder, whose etiology remains unknown, provides evidence of the effectiveness of conservative treatment approaches such as physiotherapy, analgesics, and steroid injections. Early treatment success is achieved through pain reduction and increased function rather than achieving full range of motion. Pain with movement is minimal in primary frozen shoulder in Stage 1, while night pain accompanied by activity pain is also observed in Stages 2 and 3. Secondary frozen shoulder presents with similar pain, primarily caused by inflammation in the shoulder joint capsule. Increasing range of motion without pain suppression is quite difficult in patients with frozen shoulder. Although heat or electrotherapy methods are accepted to have theoretically positive effects on pain in treatment, it is difficult to determine the effect of a single method on the natural course of the disease. For this reason, therapeutic methods are generally applied in addition to manual therapy and therapeutic exercises. Thermal tools and stretching exercises are frequently used in physiotherapy to maintain and regain flexibility. Ultrasonography, which is among the clinical diagnostic methods performed in patients with adhesive capsulitis, has shown increased thickness, especially in the coracohumeral ligament, followed by fibrous changes in the supraspinatus tendon and long head of the biceps. The effectiveness of exercise training combined with electrotherapy on many factors has been frequently investigated in the literature. However, a review of the literature did not find any studies on the effects of exercise training given in adhesive capsulitis on shoulder architecture. The fact that ultrasonographic examination, an indispensable part of the diagnosis and treatment process, provides objective data on the effects of exercise will increase the quality of the study. In this context, our study; The aim of this study is to investigate the effects of exercise training on pain, range of motion, functionality and shoulder architecture in patients with adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with adhesive capsulitis by a physician,
* Between the ages of 35-60,
* Not diagnosed with cervical disc herniation that could cause other shoulder pathologies,
* Not participating in an upper extremity-related physiotherapy program within the last 6 months,
* Volunteering individuals to participate in the study

Exclusion Criteria:

* Individuals who have undergone shoulder surgery consistent with any pathology,
* Individuals with a neurological history,
* Individuals diagnosed with diabetes mellitus (DM)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Ultrasonographic Measurement | through of the study, average 3 weeks
  Thickness and density measurements of the coracohumeral ligament, supraspinatus tendon, infraspinatus tendon, long head of biceps and deltoid fascia, which constitute the shoulder architecture of the patients and are among the structures most affected by adhesive capsulitis, will be evaluated with an Ultrasound (Measured by 7.5-10 Mhz mobile ultrasound (ALEXUS A10HRL) device.
The pain | through of the study, average 3 weeks
  Mc Gill Short Form will used to determine the type and severity of the pain. A short form of the McGill Pain Questionnaire (SF-MPQ) has been developed. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
Range of Motion | through of the study, average 3 weeks
  A Universal Goniometer will be used to assess normal range of motion. Measurements will be made regarding shoulder flexion, extension, abduction, adduction, internal and external rotation ranges of motion in three planes of the upper extremity shoulder joint, and the results will be recorded in degrees.
Upper extremity functionality | through of the study, average 3 weeks
  The Questionnaire for Arm, Shoulder, and Hand Disabilities (Q-DASH) will be used to assess individuals' upper extremity functions. This questionnaire is a self-administered measurement tool with validated validity and reliability in Turkish. The validity and reliability of the Turkish version of the DASH questionnaire (DASH-T) was conducted in Turkey by Düger et al. in 2006. The questionnaire, consisting of 30 questions, assesses the individual's ability to perform functional activities (21 items), pain (5 items), and psychosocial aspects of the disease (4 items). The total score ranges from 0 to 100, with a higher score indicating better outcomes.

SECONDARY OUTCOMES:
Kinesiophobia | through of the study, average 3 weeks
  The Tampa Kinesiophobia Scale will be used to assess the fear of movement and movement avoidance in individuals diagnosed with adhesive capsulitis. The survey, whose validity and reliability study was conducted by Yılmaz et al. in 2011, consists of 17 descriptive questions. Each question uses a 4-point Likert-type scoring system (1=Strongly disagree, 2=Agree, 3=Disagree, 4=Strongly agree). Based on the responses, the individual receives a total score between 17 and 68. A high score on the scale indicates a high degree of kinesiophobia.
The quality of Life | through of the study, average 3 weeks
  The European General Quality of Life Scale (EQ-5D) will be used to assess patients' quality of life. The EQ-5D general quality of life scale was developed in 1987 by the EuroQol group, the Western European Society for the Study of Quality of Life, and consists of two sections. The first section describes the current health profile in five subdimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Responses for each section have five options: "no problem," "mild problem," "moderate problem," "severe problem," and "extreme problem." The second section consists of a visual analog scale (VAS). In this section, individuals rate their current health status on a scale resembling a thermometer. Quality of life scores ranging from 0 to 100 are obtained from the visual analog scale. As the scale score increases, the perception of health increases in a positive direction.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yakut Y, Yakut E, Bayar K, Uygur F. Reliability and validity of the Turkish version short-form McGill pain questionnaire in patients with rheumatoid arthritis. Clin Rheumatol. 2007 Jul;26(7):1083-7. doi: 10.1007/s10067-006-0452-6. Epub 2006 Nov 15. PMID 17106618
- [Background] Do JG, Hwang JT, Yoon KJ, Lee YT. Correlation of Ultrasound Findings With Clinical Stages and Impairment in Adhesive Capsulitis of the Shoulder. Orthop J Sports Med. 2021 May 10;9(5):23259671211003675. doi: 10.1177/23259671211003675. eCollection 2021 May. PMID 33997079
- [Background] Liu J, Pan H, Bao Y, Huang L, Hu Y. The clinical utility of musculoskeletal ultrasonography in hemiplegic shoulder rehabilitation poststroke. Front Rehabil Sci. 2025 May 15;6:1576890. doi: 10.3389/fresc.2025.1576890. eCollection 2025. PMID 40443485
- [Background] Moleesaide A, Saengsuwan J, Sirasaporn P. Musculoskeletal ultrasound of the shoulder in patients with adhesive capsulitis. Biomed Rep. 2024 Oct 11;21(6):190. doi: 10.3892/br.2024.1878. eCollection 2024 Dec. PMID 39479361
- [Background] Nakano J, Yamabayashi C, Scott A, Reid WD. The effect of heat applied with stretch to increase range of motion: a systematic review. Phys Ther Sport. 2012 Aug;13(3):180-8. doi: 10.1016/j.ptsp.2011.11.003. Epub 2011 Dec 29. PMID 22814453
- [Background] Kelley MJ, Shaffer MA, Kuhn JE, Michener LA, Seitz AL, Uhl TL, Godges JJ, McClure PW. Shoulder pain and mobility deficits: adhesive capsulitis. J Orthop Sports Phys Ther. 2013 May;43(5):A1-31. doi: 10.2519/jospt.2013.0302. Epub 2013 Apr 30. No abstract available. PMID 23636125
- [Background] Kelley MJ, McClure PW, Leggin BG. Frozen shoulder: evidence and a proposed model guiding rehabilitation. J Orthop Sports Phys Ther. 2009 Feb;39(2):135-48. doi: 10.2519/jospt.2009.2916. PMID 19194024
- [Background] Hsu JE, Anakwenze OA, Warrender WJ, Abboud JA. Current review of adhesive capsulitis. J Shoulder Elbow Surg. 2011 Apr;20(3):502-14. doi: 10.1016/j.jse.2010.08.023. Epub 2010 Dec 16. No abstract available. PMID 21167743